CLINICAL TRIAL: NCT04662112
Title: Multicenter Phase I/IIa Study of NASOX (Nal-IRI + S-1 + Oxaliplatin) as First-line Treatment for Patients With Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Brief Title: Liposomal Irinotecan, S-1, and Oxaliplatin in Advanced Pancreatic Adenocarcinoma
Acronym: NASOX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NASOX
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; Liposomal irinotecan; S-1; Oxaliplatin
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NASOX (Experimental): Liposomal irinotecan+S-1+oxaliplatin
  Interventions: Drug: NASOX

INTERVENTIONS:
Drug: NASOX — Oxalipatin 60 mg/m2 IV (2 h infusion) on Day 1, every 2 weeks Nal-IRI 50-60 mg/m2 IV (FBE, 90 min infusion) on Day 1, every 2 weeks S-1 40mg/m2 oral twice daily on Day 1-7, every 2 weeks

SUMMARY:
In present study, the investigators evaluate the safety and efficacy of OIS-derived NASOX regimen (nal-IRI, S-1, oxaliplatin) in advanced pancreatic cancer. NASOX regimen contains nal-IRI, which has recently been proven effective in pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma is the seventh leading cause of cancer-related mortality worldwide, and it carries dismal prognosis with a 5-year survival rate of 1-2%. The pivotal ACCORD11 trial, FOLFIRINOX (oxaliplatin, irinotecan, 5-FU and leucovorin) has become the standard of care for patients with locally advanced or metastatic pancreatic adenocarcinoma. In daily practice, modified version of FOLFIRINOX (mFOLFIRINOX) with reduced dose of irinotecan to 150 mg/m2 and omission of bolus 5-FU has been widely used to enhance the dose intensity and safety profiles.

Despite of proven efficacy of mFOLFIRINOX in locally advanced or metastatic pancreatic cancer, further improvement in the efficacy outcomes are needed, considering that median overall survival of metastatic pancreatic cancer patients treated with FOLFIRINOX in the phase 3 trial was less than 1 year. Considering that mFOLFIRINOX often require placement of central catheterization or repeated hospitalization for continuous 5-FU infusion, novel regimens improving mFOLFIRINOX in the viewpoint of patient's quality of life is also needed. This may enhance the patient's compliance on the treatment and maximize the clinical outcomes.

Liposomal irinotecan (nal-IRI) is the novel agent enhancing the drug delivery of irinotecan and approved for the management of gemcitabine-progressed metastatic pancreatic cancer patients. Considering the hostile tumor microenvironment of pancreatic adenocarcinoma, nal-IRI may have enhanced anti-tumor activity compared to conventional irinotecan, although there are no head-to-head comparison clinical trial data, yet.

Investigators previously developed oral fluoropyrimidine-based triplet regimen (oxaliplatin, irinotecan and S-1) and investigated in 32 patients with advanced biliary tract cancer. This regimen was well tolerated and showed favorable efficacy outcome as first-line therapy with overall response rate of 50%.

In present study, investigators evaluate the safety and efficacy of OIS-derived NASOX regimen (nal-IRI, S-1, oxaliplatin) in advanced pancreatic cancer. NASOX regimen contains nal-IRI, which has recently been proven effective in pancreatic cancer. If NASOX, which is more convenient than FOLFIRINOX, proves its safety and effectiveness, it may provide an attractive alternative for pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years and older
* Histologically or cytologically confirmed, measurable pancreatic adenocarcinoma
* Treatment naïve locally advanced or metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow function as defined by platelets ≥ 100 x 109/L , neutrophils ≥ 1.5 x 109/L and hemoglobin > 9 g/dL; transfusion is allowed, provided interval is ≥ 7 days prior to screening
* Adequate renal function, with serum creatinine < 1.5 x upper limit of normal (ULN). And calculated clearance ≥ 50 mL/min/1.73m2 for patients with serum creatinine levels above or below the institutional normal value. Actual body weight should be used for calculating creatinine clearance using the Cockcroft-Gault Equation (CreatClear = Sex x ((140 - Age) / (SerumCreat)) x (Weight / 72); for patients with body mass index (BMI) >30 kg/m2, lean body weight should be used instead
* Adequate hepatic function with serum total bilirubin ≤ 2 x ULN (biliary drainage is allowed for biliary obstruction), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN is acceptable if liver metastases are present)
* History of any second malignancy in the last 3 years; patients with prior history of in-situ cancer or basal or squamous cell skin cancer are eligible. Patients with a history of other malignancies are eligible if they have been continuously disease free for at least 3 years.
* Female patients must be either surgically sterile or postmenopausal, or if of childbearing potential must have a negative pregnancy test (serum or urine) prior to enrolment and agree to use effective barrier contraception during the period of therapy and for one month after the last dose.
* Written, informed consent to the study

Exclusion Criteria:

* Endocrine or acinar pancreatic carcinoma
* Uncontrolled CNS metastases (Note: Patients who require steroids should be on a stable or decreasing dose to be eligible)
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol or a history of non-compliance
* Obstruction of gastrointestinal tract
* Active gastrointestinal bleeding
* Myocardial infarction within 6 months prior to the study medication, and other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol

  * Active infection or an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, patients with tumor fever may be enrolled), which in the investigator's opinion might compromise the patient's participation in the trial or affect the study outcome
  * Use of strong CYP3A4 inhibitors or inducers, or strong UGT1A1 inhibitors (patients are ineligible if unable to discontinue the use of strong CYP3A4 or UGT1A1 inhibitors at least 1 week or strong CYP3A4 inducers at least 2 weeks prior to receiving first dose of irinotecan liposome injection),
* presence of any contraindications for irinotecan, nal-IRI, S1 and Oxaliplatin
* Female patients who are pregnant (positive pregnancy test at screening) or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 3 weeks
Objective response rates | 6 months
  Proportion of patients with complete and partial responses defined by RECIST version 1.1

SECONDARY OUTCOMES:
Overall Survival | 1 year
  Time between study treatment and death
Progression-free survival | 1 year
  Time between study treatment and tumor progression, or death
Adverse events | 1 year
  Toxicity defined by Common Terminology Criteria version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Wainberg Z, Boland P, Lieu C, Dayyani F, Macarulla T, Zhang B, Belanger B, Moore Y, Wang T, Maxwell F, Dean A (2019) A phase 1/2, open-label, dose-expansion study of liposomal irinotecan (nal-IRI) plus 5-fluorouracil/leucovorin (5-FU/LV) and oxaliplatin (OX) in patients with previously untreated metastatic pancreatic cancer. Ann Oncol 30 Suppl 4: iv123
- [Background] Yoo C, Han B, Kim HS, Kim KP, Kim D, Jeong JH, Lee JL, Kim TW, Kim JH, Choi DR, Ha HI, Seo J, Chang HM, Ryoo BY, Zang DY. Multicenter Phase II Study of Oxaliplatin, Irinotecan, and S-1 as First-line Treatment for Patients with Recurrent or Metastatic Biliary Tract Cancer. Cancer Res Treat. 2018 Oct;50(4):1324-1330. doi: 10.4143/crt.2017.526. Epub 2018 Jan 8. PMID 29334603
- [Background] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328